CLINICAL TRIAL: NCT03754452
Title: Evaluation of the Prevalence, the Diagnosis Tests, and the Associated Morbimortality of Sarcopenia in Hepatobiliary Surgery
Brief Title: Evaluation of the Sarcopenia in Hepatobiliary Surgery
Acronym: SARFO
Status: Terminated | Type: Observational
Why Stopped: No inclusion
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-A1104-51
Record Dates: First submitted 2018-11-12; First posted 2018-11-27 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sarcopenia; Hepatobiliary Disease; Postoperative Complications; Surgery
MeSH Terms: conditions — Sarcopenia; Digestive System Diseases; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The sarcopenia is defined as a loss of muscle mass and a loss of muscle function ( strength or performance). Some studies showed that the sarcopenia increase the postoperative complications and the overall survival in abdominal surgery. But the sarcopenia is not evaluated in the Hepatobiliary surgery. This prospective, monconcentrique study aim to evaluate the prevalence of sarcopenia, and its associated morbimortality in hepatobiliary surgery for malignant or benign tumors.

ELIGIBILITY:
Inclusion Criteria:

* hepatobiliary surgery
* scheduled surgery
* oral consent

Exclusion Criteria:

* pregnancy
* patient under low protection
* emergency surgery
* hepatic encephalopathy stage II, III and IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - all patients who should have a hepatobiliary surgery for malignant and benign tumor in the universitary hospital center of Angers
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
the number of patients with a sarcopenia before having a hepatobiliary surgery mesured by impedancemetry and by the muscular force or the speed walking | 1 month
  for the man : i/impedancemetry BMI<8,87kg/m2 and ii/ a muscular force < 30kg or a walking speed <0,8m/s
the number of patients with a sarcopenia before having a hepatobiliary surgery mesured by impedancemetry and by the muscular force or the speed walking | 1 month
  for the woman: i/impedancemetry BMI<6,42kg/m2 and ii/muscular force < 20kg or a walking speed <0,8m/s

SECONDARY OUTCOMES:
comparison between the impedancemetry and the abdominopevis CT for the diagnosis of sarcopenia | 3 months
  * impedancemetry used to evaluate the muscular mass
  * abdominopelvis CT evualate the muscular mass by measuring the muscular area on the L3 section
comparison of the postoperatives complications using the clavien dindo classsification between the patient with sarcopenia and the patient without sarcopenia. | 4 months
  postoperatives complications evualuated according the clavien dindo classification are : death, nausea, vomit, need of nasogastric tube, liver failure with jaundice, ascites, liver encephalopathy, biliary fistula, biliary peritonitis, hernia, parietal abcess, urinary infection, urinary retention, hematoma, pulmonary embolism, pulmonary infection, pleural effusion, atelectasis, renal failure, hyponatremia, hypernatremia, hypokaliema, hyperkaliema the post operative complication evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Julien BARBIEUX, Dr, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No